CLINICAL TRIAL: NCT01651780
Title: Effect of Bivalirudin on Aortic Valve Intervention Outcomes 2/3 (BRAVO 2/3)
Brief Title: Open-label, Randomized Trial in Participants Undergoing TAVR to Determine Safety & Efficacy of Bivalirudin vs UFH
Acronym: BRAVO 2/3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Medicines Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TMC-BIV-11-02; 2012-000632-26 (EudraCT Number)
Record Dates: First submitted 2012-07-24; First posted 2012-07-27 (Estimated); Results first posted 2017-02-27 (Actual); Last update posted 2017-04-07 (Actual); Status verified 2017-03

CONDITIONS: Severe Aortic Stenosis; Transcatheter Aortic Valve Replacement; Aortic Valve Replacement
Keywords: Transcatheter aortic valve replacement; Aortic valve replacement; Severe aortic stenosis
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — bivalirudin; Heparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | US Export: Yes

ARMS (2):
- Bivalirudin (Experimental): Bivalirudin administered as a bolus and intravenous (IV) infusion during TAVR. It was recommended that the bolus (0.75 milligrams per kilogram [mg/kg]) be directly administered through the valve delivery sheath immediately following its successful delivery via percutaneous femoral access. Systemic IV administration of the bolus dose was also acceptable. The bivalirudin IV infusion was initiated immediately after the bolus administration. All wires, catheters, and sheaths were to be flushed with heparinized saline.
  Interventions: Drug: Bivalirudin
- Unfractionated heparin (UFH) (Active Comparator): The dose of UFH adhered to the standard institutional practice. An activated clotting time (ACT) target ≥250 seconds was recommended. All wires, catheters, and sheaths were to be flushed with heparinized saline.
  Interventions: Drug: Unfractionated Heparin

INTERVENTIONS:
Drug: Bivalirudin — Bivalirudin is an anticoagulant that binds directly to thrombin in a bivalent and reversible fashion.
  Other Names: AngioMAX; Angiox
  Arms: Bivalirudin
Drug: Unfractionated Heparin — Unfractionated heparin is an anticoagulant.
  Other Names: Heparin
  Arms: Unfractionated heparin (UFH)

SUMMARY:
The objective of this study is to assess the safety and efficacy of using bivalirudin instead of unfractionated heparin (UFH) in transcatheter aortic valve replacements (TAVR). The primary hypothesis of BRAVO 3 was that bivalirudin would reduce major bleeding compared with heparin in TAVR procedures. Results for all participants enrolled into the randomized trial (BRAVO 3) are presented.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, ≥18 years of age
* High risk (Euroscore ≥18, or considered inoperable) for surgical aortic valve replacement
* Undergoing TAVR via transfemoral arterial access
* Provide written informed consent before initiation of any study related procedures

Exclusion Criteria:

* Any known contra-indication to the use of bivalirudin (except presence of severe renal impairment [glomerular filtration rate (GFR) <30 milliliters (mL)/minute] since these participants will be included in the trial or UFH
* Refusal to receive blood transfusion
* Mechanical valve (any location) or mitral bioprosthetic valve
* Extensive calcification of the common femoral artery, or minimal luminal diameter <6.5 millimeters (mm)
* Use of elective surgical cut-down for transfemoral access
* Concurrent performance of percutaneous coronary intervention with TAVR
* International normalized ratio (INR) ≥2 on the day of TAVR procedure or known history of bleeding diathesis
* History of hemorrhagic stroke, intracranial hemorrhage, intracerebral mass or aneurysm, or arteriovenous malformation
* Severe left ventricular dysfunction (left ventricular ejection fraction <15%)
* Severe aortic regurgitation or mitral regurgitation (4+)
* Hemodynamic instability (for example, requiring inotropic or intra-aortic balloon pump support) within 2 hours of the procedure
* Dialysis dependent
* Administration of thrombolytics, glycoprotein IIb/IIIa inhibitors, or warfarin in the 3 days prior to the procedure
* Acute myocardial infarction, major surgery, or any therapeutic cardiac procedure (other than balloon aortic valvuloplasty) within 30 days
* Percutaneous coronary intervention within 30 days
* Upper gastrointestinal or genitourinary bleed within 30 days
* Stroke or transient ischemic attack within 30 days
* Any surgery or biopsy within 2 weeks
* Administration of:

  * UFH within 30 minutes of the procedure
  * Enoxaparin within 8 hours of the procedure
  * Fondaparinux or other low-molecular-weight heparins (LMWHs) within 24 hours of the procedure
  * Dabigatran, rivaroxaban, or other oral anti-Xa or antithrombin agent within 48 hours of the procedure
  * Thrombolytics, glycoprotein IIb/IIIa inhibitor, or warfarin within 72 hours of the procedure
* Absolute contraindications or allergy that cannot be pre-medicated to iodinated contrast
* Contraindications or allergy to aspirin or clopidogrel
* Known or suspected pregnant women or nursing mothers. Women of child-bearing potential will be asked if they are pregnant and will be tested for pregnancy
* Previous enrollment in this study
* Treatment with other investigational drugs or devices within the 30 days preceding enrollment or planned use of other investigational drugs or devices before the primary endpoint of this study has been reached

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 803 (Actual)
Dates: Start 2012-10; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thierry Lefevre, MD, Principal Investigator — Hôpital Privé Jacques Cartier; Eberhardt Grube, MD, Principal Investigator — University Hospital, Bonn; George D Dangas, MD, PhD, Study Director — The Zena and Michael A. Wiener Cardiovascular Institute; Prodromos Anthopoulos, MD, Study Director — The Medicines Company
Locations (33):
- Canada (2):
  - Montreal Heart Institute, Montreal, Quebec
  - St. Paul´s Hospital Providence Health Care, Vancouver
- France (7):
  - Clinique Pasteur, Unité de Cardiologie Interventionnelle, Toulouse, Cedex 3
  - CHU de Toulouse, Toulouse, Cedex 9
  - CHU Jean Minjoz, Service de Cardiologie, Besançon
  - Centre Hospitalier de Lyon, Bron
  - Department of Cardiology, CHRU Lille, Lille
  - Institut Hospitalier Jacques Cartier, Massy
  - Service de Cardiologie, Centre Hospitalo-Universitaire, Hôpital Charles-Nicolle, Rouen
- Germany (13):
  - University Heart Centre, Clinic of Inner Medicine 1 Cardiology, Jena, Lobeda Ost
  - Universitätsklinikum Bonn, Bonn
  - Klinikum links der Weser Bremen, Bremen
  - Elisabeth-Krankenhaus Essen, Essen
  - Freiburg University, Freiburg im Breisgau
  - Asklepios St. Georg Hamburg, Hamburg
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Universität Leipzig - Herzzentrum GmbH, Leipzig
  - Universitätsmedizin der Johannes Gutenberg-Universitat Mainz, Mainz
  - LMU Munich, Klinikum der Universität München, Munich
  - Deutsches Herzzentrum München, München
  - Helios Heart Center Siegburg, Siegburg
- Italy (5):
  - Ferraroto Hospital, University of Catania, Catania
  - Ospedale San Raffaele U.O. Cardiologia Interventistica, Milan
  - Azienda Ospedaliero-Universitaria Pisana, Pisa
  - Azienda Ospedaliera San Camillo-Forlanini, Roma
  - Policlinico Umberto I, Università La Sapienza, Roma
- Netherlands (2):
  - St. Antonius Ziekenhuis, Nieuwegein
  - University Medical Center Utrecht, Utrecht
- Switzerland (2):
  - Cardiology University Hospital Basel, Basel
  - Universitätsklinik Bern, Bern
- United Kingdom (2):
  - The Royal Sussex County Hospital, Brighton, East Sussex
  - Hammersmith Hospital, London

REFERENCES:
- [Derived] Van Belle E, Hengstenberg C, Lefevre T, Kupatt C, Debry N, Husser O, Pontana F, Kuchcinski G, Deliargyris EN, Mehran R, Bernstein D, Anthopoulos P, Dangas GD; BRAVO-3 MRI Study Investigators. Cerebral Embolism During Transcatheter Aortic Valve Replacement: The BRAVO-3 MRI Study. J Am Coll Cardiol. 2016 Aug 9;68(6):589-599. doi: 10.1016/j.jacc.2016.05.006. Epub 2016 May 18. PMID 27208464
- [Derived] Dangas GD, Lefevre T, Kupatt C, Tchetche D, Schafer U, Dumonteil N, Webb JG, Colombo A, Windecker S, Ten Berg JM, Hildick-Smith D, Mehran R, Boekstegers P, Linke A, Tron C, Van Belle E, Asgar AW, Fach A, Jeger R, Sardella G, Hink HU, Husser O, Grube E, Deliargyris EN, Lechthaler I, Bernstein D, Wijngaard P, Anthopoulos P, Hengstenberg C; BRAVO-3 Investigators. Bivalirudin Versus Heparin Anticoagulation in Transcatheter Aortic Valve Replacement: The Randomized BRAVO-3 Trial. J Am Coll Cardiol. 2015 Dec 29;66(25):2860-2868. doi: 10.1016/j.jacc.2015.10.003. Epub 2015 Oct 15. PMID 26477635

RESULTS

PARTICIPANT FLOW:
Groups:
- Bivalirudin: Bivalirudin administered as a bolus and intravenous (IV) infusion during transcatheter aortic valve replacement (TAVR). It was recommended that the bolus (0.75 milligrams per kilogram [mg/kg]) be directly administered through the valve delivery sheath immediately following its successful delivery via percutaneous femoral access. Systemic IV administration of the bolus dose was also acceptable. The bivalirudin IV infusion was initiated immediately after the bolus administration. All wires, catheters, and sheaths were to be flushed with heparinized saline.
Period: Overall Study
Arm/Group | Bivalirudin | Unfractionated Heparin (UFH)
Started | 405 | 398
Intent-To-Treat (ITT) Population | 404 | 398
Received at Least 1 Dose of Study Drug | 393 (All but 1 participant in the bivalirudin group (withdrew consent) comprised the ITT population.) | 394
BRAVO 2 Feasibility Cohort | 65 (1st 2 participants/site made up the bivalirudin feasibility cohort (BRAVO2) and analyzed separately.) | 0 (1st 2 participants/site made up the bivalirudin feasibility cohort (BRAVO2) and analyzed separately.)
Completed | 394 | 388
Not Completed | 11 | 10
Not completed — Physician decision: No 30-day visit | 2 | 1
Not completed — Reason Not Specified: No 30-day visit | 2 | 2
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Inclusion/Exclusion Criteria Not Met | 3 | 0
Not completed — Lost to Follow-up | 1 | 2
Not completed — Physician decision: Day 30 visit <23 day | 1 | 5

BASELINE CHARACTERISTICS:
Population: Participants in the ITT population.
Groups:
- Unfractionated Heparin (UFH): The dose of UFH adhered to the standard institutional practice. An ACT target ≥250 seconds was recommended. All wires, catheters, and sheaths were to be flushed with heparinized saline.
- Total: Total of all reporting groups
Arm/Group | Bivalirudin | Unfractionated Heparin (UFH) | Total
Number analyzed (Participants) | 404 | 398 | 802
Age, Continuous [Mean (Standard Deviation); unit: years] | 82.3 (6.5) | 82.3 (6.5) | 82.3 (6.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 195 | 196 | 391
  Male | 209 | 202 | 411
Region of Enrollment [Number; unit: participants]
  Canada | 36 | 38 | 74
  Netherlands | 10 | 10 | 20
  Italy | 37 | 39 | 76
  United Kingdom | 8 | 10 | 18
  France | 108 | 106 | 214
  Switzerland | 25 | 22 | 47
  Germany | 180 | 173 | 353

OUTCOME MEASURES:

1. Primary Outcome: Major Bleeding (BARC ≥3b) at 48 Hours or Before Hospital Discharge
Description: Major bleeding (Bleeding Academic Research Consortium [BARC] type ≥3b) was defined as follows:
  * Bleeds that were evident clinically, or by laboratory or imaging results, which resulted in surgical intervention or administration of IV vasoactive drugs; overt bleeds with a hemoglobin drop of at least 5 grams per deciliter (g/dL); and bleeding that caused cardiac tamponade.
  * BARC 3c includes intracranial or intraocular bleeds that compromised vision.
  * BARC type 4 (Coronary Artery Bypass Grafting [CABG]-related bleeding) includes perioperative intracranial bleeding within 48 hours, bleeds that result in reoperation following closure of sternotomy for the purpose of controlling bleeding, bleeds that result in treatment with transfusion of ≥5 units of whole blood or packed red blood cells within a 48 hour period; and chest tube output ≥2 liters (L) within a 24-hour period.
  * BARC type 5, fatal bleeding, describes bleeds that directly result in death with no other cause.
Time Frame: at 48 hours or discharge, whichever occurs first
Population: Participants in the ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Bivalirudin | Unfractionated Heparin (UFH)
Number analyzed (Participants) | 404 | 398
percentage of participants | 6.9 | 9
Statistical Analysis 1: Comparison: Bivalirudin vs Unfractionated Heparin (UFH); Test type: Non-Inferiority or Equivalence — If non-inferiority was confirmed, then superiority analysis was pursued; p = 0.2692, Chi-squared; Relative Risk = 0.77, 95% CI 2-sided [0.48 to 1.23]

2. Primary Outcome: Net Adverse Clinical Events (NACE) at up to 30 Days
Description: The net adverse cardiac events (NACE) at 30 days is the composite of major adverse cardiovascular events (MACE) + major bleeding (BARC type ≥3b). The composite of MACE is defined as all-cause mortality, myocardial infarction (MI), and stroke. A participant was defined to have a composite event if the participant experienced at least 1 of the components. If the participant did not have any of the components, then he or she did not have the composite endpoint. If a participant had more than 1 of the components, he or she was only counted once in the determination of the total number of participants experiencing the composite endpoint.
Time Frame: up to 30 days after procedure
Population: Participants in the ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Bivalirudin | Unfractionated Heparin (UFH)
Number analyzed (Participants) | 404 | 398
percentage of participants | 14.4 | 16.1
Statistical Analysis 1: Comparison: Bivalirudin vs Unfractionated Heparin (UFH); Test type: Non-Inferiority or Equivalence — If non-inferiority was confirmed, then superiority analysis was pursued; p = 0.4967, Chi-squared; Relative Risk = 0.89, 95% CI 2-sided [0.64 to 1.24]

3. Secondary Outcome: NACE at 48 Hours or Before Hospital Discharge
Description: NACE at 48 hours or before hospital discharge is the composite of major adverse cardiovascular events (MACE) + major bleeding (BARC type ≥3b). The composite of MACE is defined as all-cause mortality, MI, and stroke. A participant was defined to have a composite event if the participant experienced at least 1 of the components. If the participant did not have any of the components, then he or she did not have the composite endpoint. If a participant had more than 1 of the components, he or she was only counted once in the determination of the total number of participants experiencing the composite endpoint.
Time Frame: at 48 hours or before hospital discharge, whichever occurred earlier
Population: Participants in the ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Bivalirudin | Unfractionated Heparin (UFH)
Number analyzed (Participants) | 404 | 398
percentage of participants | 8.9 | 12.6

4. Secondary Outcome: Major Adverse Cardiac Events (MACE) Including Death, Non-fatal MI, and Stroke
Description: The percentage of participants reporting a MACE overall and the individual components of MACE (including death, non-fatal MI, and stroke) are presented.
Time Frame: at 48 hours or before hospital discharge, whichever occurred earlier, and at up to 30 days (±7 days)
Population: Participants in the ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Bivalirudin | Unfractionated Heparin (UFH)
Number analyzed (Participants) | 404 | 398
percentage of participants
  MACE at 48 hours or before hospital discharge | 3.5 | 4.8
  Death at 48 hours or before hospital discharge | 1.5 | 1.8
  MI at 48 hours or before hospital discharge | 0 | 1.3
  Stroke at 48 hours or before hospital discharge | 2 | 2
  MACE at up to 30 days | 7.7 | 8
  Death at up to 30 days | 4.7 | 4.8
  MI at up to 30 days | 0.5 | 1.8
  Stroke at up to 30 days | 3.5 | 2.8

5. Secondary Outcome: Major Bleeding According to Additional Scales (VARC, TIMI, GUSTO, ACUITY/HORIZONS)
Description: Percentage of participants with major bleeding according to the following scales:
  * Valve Academic Research Consortium (VARC)=life threatening, disabling bleeding, or major bleeding
  * Thrombolysis in Myocardial Infarction (TIMI)=major bleeding
  * Global Use of Strategies to Open Occluded Coronary Arteries (GUSTO)=severe or moderate
  * Acute Catheterization and Urgent Intervention Triage StrategY (ACUITY)/Harmonizing Outcomes with RevasculariZatiON and Stents (HORIZONS)=major bleeding
Time Frame: at 48 hours or hospital discharge, whichever occurred earlier, and at up to 30 days (±7 days) follow-up
Population: Participants in the ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Bivalirudin | Unfractionated Heparin (UFH)
Number analyzed (Participants) | 404 | 398
percentage of participants
  VARC at 48 hours or before hospital | 21.8 | 19.6
  TIMI at 48 hours or before hospital | 4 | 6.5
  GUSTO at 48 hours or hospital discharge | 13.9 | 11.6
  ACUITY/HORIZONS at 48 hours or hospital discharge | 26 | 24.4
  VARC at 30 days | 26.5 | 24.6
  TIMI at 30 days | 5.7 | 7.3
  GUSTO at 30 days | 16.3 | 14.6
  ACUITY/HORIZONS at 30 days | 33.4 | 29.6

6. Secondary Outcome: Transient Ischemic Attack
Description: The percentage of participants reporting transient ischemic attack is presented.
Time Frame: at 48 hours or before hospital discharge, whichever occurred earlier, and at up to 30 days (±7 days)
Population: Participants in the ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Bivalirudin | Unfractionated Heparin (UFH)
Number analyzed (Participants) | 404 | 398
percentage of participants
  at 48 hours or before hospital discharge | 0 | 0
  at up to 30 days (±7 days) follow-up | 0 | 0

7. Secondary Outcome: Acute Kidney Injury
Description: The percentage of participants reporting acute kidney injury is presented.
Time Frame: at 48 hours or hospital discharge, whichever occurred earlier, and at up to 30 days (±7 days) follow-up
Population: Participants in the ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Bivalirudin | Unfractionated Heparin (UFH)
Number analyzed (Participants) | 404 | 398
percentage of participants
  at 48 hours or before hospital discharge | 10.9 | 6.5
  at up to 30 days (±7 days) follow-up | 18.8 | 13.8

8. Secondary Outcome: Major Vascular Complications
Description: The percentage of participants reporting a major vascular complications as defined by VARC is presented.
Time Frame: at 48 hours or before hospital discharge, whichever occurred earlier, and at up to 30 days (±7 days)
Population: Participants in the ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Bivalirudin | Unfractionated Heparin (UFH)
Number analyzed (Participants) | 404 | 398
percentage of participants
  at 48 hours or before hospital discharge | 8.7 | 9
  at up to 30 days (±7 days) follow-up | 9.2 | 9.5

9. Secondary Outcome: Acquired Thrombocytopenia
Description: The percentage of participants reporting acquired thrombocytopenia is presented.
Time Frame: at 48 hours or before hospital discharge, whichever occurred earlier, and at up to 30 days (±7 days)
Population: Participants in the ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Bivalirudin | Unfractionated Heparin (UFH)
Number analyzed (Participants) | 404 | 398
percentage of participants
  at 48 hours or before hospital discharge | 16.6 | 17.3
  at up to 30 days (±7 days) | 24 | 23.1

10. Secondary Outcome: New Onset Atrial Fibrillation/Flutter
Description: The percentage of participants reporting new onset atrial fibrillation/flutter is presented.
Time Frame: at 48 hours or before hospital discharge, whichever occurred earlier, and at up to 30 days (±7 days)
Population: Participants in the ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Bivalirudin | Unfractionated Heparin (UFH)
Number analyzed (Participants) | 404 | 398
percentage of participants
  at 48 hours or before hospital discharge | 3.2 | 2.5
  at up to 30 days (±7 days) follow-up | 5.4 | 4

11. Secondary Outcome: Timing Effect on Bleeding Event Rate up to 48 Hours or Hospital Discharge
Description: The effect of timing on bleeding event rates (the percentage of participants with an incidence of major bleeding) is presented.
Time Frame: Up to 48 hours after procedure or at hospital discharge (but also includes any subsequent hospitalizations)
Population: Participants in the ITT population with an incidence of major bleeding. Participants were categorized as "First half of study site's enrolled participants" (Bivalirudin, N=173; UFH, N=173) and "Second half of study site's enrolled participants" (Bivalirudin, N=171; UFH, N=165). Only sites with >20 participants are included in this analysis.
Measure: Number; unit: percentage of participants
Groups:
- Bivalirudin: First Half of Study Site's Enrolled Participants: Bivalirudin administered as a bolus and intravenous (IV) infusion during TAVR. It was recommended that the bolus (0.75 milligrams per kilogram [mg/kg]) be directly administered through the valve delivery sheath immediately following its successful delivery via percutaneous femoral access. Systemic IV administration of the bolus dose was also acceptable. The bivalirudin IV infusion was initiated immediately after the bolus administration. All wires, catheters, and sheaths were to be flushed with heparinized saline. This includes the first half of the site's enrolled participants, and only sites with more than 20 participants are included in this analysis.
- Bivalirudin: Second Half of Study Site's Enrolled Participants: Bivalirudin administered as a bolus and intravenous (IV) infusion during TAVR. It was recommended that the bolus (0.75 milligrams per kilogram [mg/kg]) be directly administered through the valve delivery sheath immediately following its successful delivery via percutaneous femoral access. Systemic IV administration of the bolus dose was also acceptable. The bivalirudin IV infusion was initiated immediately after the bolus administration. All wires, catheters, and sheaths were to be flushed with heparinized saline. This includes the second half of the site's enrolled participants, and only sites with more than 20 participants are included in this analysis.
- UFH: First Half of Study Site's Enrolled Participants: The dose of UFH adhered to the standard institutional practice. An ACT target ≥250 seconds was recommended. All wires, catheters, and sheaths were to be flushed with heparinized saline. This includes the first half of the site's enrolled participants, and only sites with more than 20 participants are included in this analysis.
- UFH: Second Half of Study Site's Enrolled Participants: The dose of UFH adhered to the standard institutional practice. An ACT target ≥250 seconds was recommended. All wires, catheters, and sheaths were to be flushed with heparinized saline. This includes the second half of the site's enrolled participants, and only sites with more than 20 participants are included in this analysis.
Arm/Group | Bivalirudin: First Half of Study Site's Enrolled Participants | Bivalirudin: Second Half of Study Site's Enrolled Participants | UFH: First Half of Study Site's Enrolled Participants | UFH: Second Half of Study Site's Enrolled Participants
Number analyzed (Participants) | 173 | 171 | 173 | 165
percentage of participants | 6.4 | 6.4 | 11.6 | 8.5

12. Secondary Outcome: Bleeding BARC 3a, BARC Types 1 or 2, and TIMI Minor
Description: The percentage of participants with moderate bleeding as defined by BARC 3a and minor bleeding as defined as BARC type 1 and 2 and TIMI minor is presented.
Time Frame: at 48 hours or hospital discharge, whichever occurred earlier, and at up to 30 days (±7 days) follow-up
Population: Participants in the ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Bivalirudin | Unfractionated Heparin (UFH)
Number analyzed (Participants) | 404 | 398
percentage of participants
  BARC 3a at 48 hours or hospital discharge | 15.6 | 13.3
  BARC types 1 and 2 at 48 hours or discharge | 20.8 | 21.1
  TIMI minor at 48 hours or hospital discharge | 16.6 | 14.3
  BARC 3a at 30 days | 18.8 | 17.3
  BARC types 1 and 2 at 30 days | 27.7 | 25.6
  TIMI minor at 30 days | 21.3 | 19.3

ADVERSE EVENTS:
Arm/Group | Bivalirudin | Unfractionated Heparin (UFH)
Serious Adverse Events (participants affected / at risk) | 112/393 | 116/394
Other Adverse Events (participants affected / at risk) | 73/393 | 70/394
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bivalirudin (N=393) | Unfractionated Heparin (UFH) (N=394)
Hypotension (Vascular disorders) | 2 | 1
Peripheral ischaemia (Vascular disorders) | 0 | 2
Aortic dissection (Vascular disorders) | 1 | 0
Circulatory collapse (Vascular disorders) | 1 | 0
Femoral artery dissection (Vascular disorders) | 1 | 0
Haemodynamic instability (Vascular disorders) | 0 | 1
Hypertensive crisis (Vascular disorders) | 0 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 0
Peripheral artery thrombosis (Vascular disorders) | 1 | 0
Phlebitis (Vascular disorders) | 1 | 0
Shock (Vascular disorders) | 0 | 1
Intestinal anastomosis (Surgical and medical procedures) | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Anaphylactic shock (Immune system disorders) | 1 | 0
Death (General disorders) | 1 | 1 — Organ system includes administration site conditions.
Device leakage (General disorders) | 1 | 1 — Organ system includes administration site conditions.
Thrombosis in device (General disorders) | 2 | 0 — Organ system includes administration site conditions.
Device dislocation (General disorders) | 0 | 1 — Organ system includes administration site conditions.
General physical health deterioration (General disorders) | 1 | 0 — Organ system includes administration site conditions.
Hyperthermia (General disorders) | 1 | 0 — Organ system includes administration site conditions.
Multi-organ failure (General disorders) | 0 | 1 — Organ system includes administration site conditions.
Non-cardiac chest pain (General disorders) | 1 | 0 — Organ system includes administration site conditions.
Pyrexia (General disorders) | 1 | 0 — Organ system includes administration site conditions.
Sudden death (General disorders) | 1 | 0 — Organ system includes administration site conditions.
Confusional state (Psychiatric disorders) | 1 | 0
Panic attack (Psychiatric disorders) | 0 | 1
Cardiac valve replacement (Injury, poisoning and procedural complications) | 3 | 0
Cardiac valve rupture (Injury, poisoning and procedural complications) | 0 | 2
Fall (Injury, poisoning and procedural complications) | 0 | 2
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 1 | 0
Vascular procedure complication (Injury, poisoning and procedural complications) | 1 | 0
Atrioventricular block complete (Cardiac disorders) | 46 | 34
Bundle branch block left (Cardiac disorders) | 7 | 10
Bradycardia (Cardiac disorders) | 2 | 7
Cardiac arrest (Cardiac disorders) | 2 | 7
Atrioventricular block second degree (Cardiac disorders) | 2 | 6
Atrioventricular block first degree (Cardiac disorders) | 3 | 4
Atrioventricular block (Cardiac disorders) | 2 | 4
Ventricular tachycardia (Cardiac disorders) | 4 | 1
Cardiac failure acute (Cardiac disorders) | 1 | 3
Aortic valve incompetence (Cardiac disorders) | 1 | 1
Cardiac tamponade (Cardiac disorders) | 1 | 1
Cardiogenic shock (Cardiac disorders) | 0 | 2
Coronary artery occlusion (Cardiac disorders) | 0 | 2
Ventricular fibrillation (Cardiac disorders) | 1 | 1
Ventricular tachyarrhythmia (Cardiac disorders) | 1 | 1
Bifascicular block (Cardiac disorders) | 1 | 0
Bradyarrhythmia (Cardiac disorders) | 1 | 0
Cardiac perforation (Cardiac disorders) | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0
Cardiopulmonary failure (Cardiac disorders) | 1 | 0
Coronary artery stenosis (Cardiac disorders) | 0 | 1
Ischaemic cardiomyopathy (Cardiac disorders) | 0 | 1
Low cardiac output syndrome (Cardiac disorders) | 0 | 1
Pericardial effusion (Cardiac disorders) | 1 | 0
Sick sinus syndrome (Cardiac disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Bundle branch block (Cardiac disorders) | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Chronic obstructive pulmonary (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 3 | 0
Carotid artery stenosis (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Cognitive disorder (Nervous system disorders) | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 0 | 1
Haemorrhagic stroke (Nervous system disorders) | 1 | 0
Loss of consciousness (Nervous system disorders) | 0 | 1
Myasthenia gravis (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 1 | 1
Abdominal hernia (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1
Intestinal infarction (Gastrointestinal disorders) | 0 | 1
Intestinal ischaemia (Gastrointestinal disorders) | 1 | 0
Umbilical hernia, obstructive (Gastrointestinal disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 2
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Pneumonia (Infections and infestations) | 2 | 2
Bronchopneumonia (Infections and infestations) | 0 | 2
Sepsis (Infections and infestations) | 1 | 1
Bronchitis (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 0 | 1
Intervertebral discitis (Infections and infestations) | 1 | 0
Klebsiella infection (Infections and infestations) | 0 | 1
Pneumonia viral (Infections and infestations) | 1 | 0
Postoperative wound infection (Infections and infestations) | 0 | 1
Pseudomonas infection (Infections and infestations) | 1 | 0
Septic encephalopathy (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
Cardiac failure (Cardiac disorders) | 6 | 10
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bivalirudin (N=393) | Unfractionated Heparin (UFH) (N=394)
Hypertension (Vascular disorders) | 19 | 16
Bundle branch block left (Cardiac disorders) | 15 | 16
Pyrexia (General disorders) | 12 | 19 — Organ system includes administration site conditions.
Confusional state (Psychiatric disorders) | 14 | 10
Back pain (Musculoskeletal and connective tissue disorders) | 13 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No